CLINICAL TRIAL: NCT06771102
Title: Performance Characteristics and Technical Outcomes of Single-use Gastroscopes Used Bedside Versus Reusable Gastroscopes Used in the Endoscopy Unit Evaluated in Subacute Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Camilla Kjelkvist-Born, Principal Investigator, Zealand University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUSUES_bedsideGAS
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Upper Gastrointestinal Disorder
Keywords: Gastroscopy; Upper endoscopy; Gastroscope; Single-use; Reusable; Bedside
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, quality assurance study. Non-randomized, controlled single center feasibility study. Comparing a period where subacute gastroscopies are performed in the endoscopy unit (reusable gastroscopes) with a period where they are performed bedside in the patients room (single-use gastroscopes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reusable gastroscope in the endoscopy unit (Active Comparator): In the first period the subacute gastroscopies will be performed with a reusable gastroscope in the endoscopy unit.
  Interventions: Device: Diagnostic gastroscopes, Olympus
- Single-use gastroscope bedside in the patient's room (Experimental): In the second period the subacute gastroscopies will be performed with a reusable gastroscope in bedside in the patients' rooms.
  Interventions: Device: Ambu aScope Gastro

INTERVENTIONS:
Device: Ambu aScope Gastro — CE-marked single-use gastroscopes from Ambu are used in the single-use group.
  Arms: Single-use gastroscope bedside in the patient's room
Device: Diagnostic gastroscopes, Olympus — Reusable gastroscopes from Olympus are used in the reusable group.
  Arms: Reusable gastroscope in the endoscopy unit

SUMMARY:
The aim of this study is to investigate whether single-use gastroscopes used bedside can reduce the time from indication to procedure compared with re-usable gastroscopes used at the endoscopy unit in patients referred to a subacute gastroscopy.

Participants in the first period will be scheduled for gastroscopy with a re-usable gastroscope in the endoscopy unit, whereas participants during the second period will have a gastroscopy performed at the ward (bed-side) with a single-use gastroscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender, 18 years of age or older admitted to the acute section of the surgical department (Kir2) at Zealand University Hospital referred to early EGD without general anesthesia.

Exclusion Criteria:

* ASA-score of 4 or higher
* Unstable patient
* Suspicion of ventricular retention
* Suspicion of active bleeders
* Need for expert endoscopist to perform the procedure, e.g. stenting
* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Time from the indication/decision for early endoscopy to procedure | From indication to procedure, up to two weeks

SECONDARY OUTCOMES:
Time from indication to the discharge | From indication to discharge, up to 3 months
Time from procedure to discharge | From procedure to discharge, up to 3 months
Duration of the procedure | During the procedure
Did the patient need sedation or local anesthetic throat spray | During the procedure
Technical success | From admission to discharge, up to 3 months
  Technical success is defined as the ability to complete the procedure adequately based on the indication and guidelines.
Sufficient ability to target the biopsy if taken | During the procedure
  Successful biopsy that provides the pathologist with sufficient material to either confirm or rule out a diagnosis. If the biopsy is inadequate, the pathologist will note this in the report.
Complications to gastroscopy | 24 and 72 hour follow-up after procedure
30th day mortality | 30 days
Readmission | 30 days after procedure
  Does the patient need readmission after discharge?
The necessity for a new gastroscopy, including the reasons justifying it | During admission, up to 3 months
  Did the patient need a new gastroscopy during admission? If so, what is the reason for that, according to the patient's medical record?
Endoscopists' rating of the gastroscope | Right after procedure
  The endoscopist's rating of the gastroscope
Learning curve for nurses at the surgical department | During the second period (one year)
  Following each procedure, the nurses will complete a short questionnaire evaluating their level of comfort (from 1-5) during the various steps of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Bremholm Hansen, PhD, ass.prof, Study Chair — Surgical department of Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez de Santiago E, Dinis-Ribeiro M, Pohl H, Agrawal D, Arvanitakis M, Baddeley R, Bak E, Bhandari P, Bretthauer M, Burga P, Donnelly L, Eickhoff A, Hayee B, Kaminski MF, Karlovic K, Lorenzo-Zuniga V, Pellise M, Pioche M, Siau K, Siersema PD, Stableforth W, Tham TC, Triantafyllou K, Tringali A, Veitch A, Voiosu AM, Webster GJ, Vienne A, Beilenhoff U, Bisschops R, Hassan C, Gralnek IM, Messmann H. Reducing the environmental footprint of gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) and European Society of Gastroenterology and Endoscopy Nurses and Associates (ESGENA) Position Statement. Endoscopy. 2022 Aug;54(8):797-826. doi: 10.1055/a-1859-3726. Epub 2022 Jul 8. PMID 35803275
- [Background] Namburar S, von Renteln D, Damianos J, Bradish L, Barrett J, Aguilera-Fish A, Cushman-Roisin B, Pohl H. Estimating the environmental impact of disposable endoscopic equipment and endoscopes. Gut. 2022 Jul;71(7):1326-1331. doi: 10.1136/gutjnl-2021-324729. Epub 2021 Dec 1. PMID 34853058
- [Background] Le NNT, Hernandez LV, Vakil N, Guda N, Patnode C, Jolliet O. Environmental and health outcomes of single-use versus reusable duodenoscopes. Gastrointest Endosc. 2022 Dec;96(6):1002-1008. doi: 10.1016/j.gie.2022.06.014. Epub 2022 Jun 17. PMID 35718068
- [Background] Cennamo V, Botter A, Landi S, Graziosi F, Bassi M, Dabizzi E, Ghersi S, Cerone G, Bonfiglioli R. Can single-use versus standard duodenoscope improve ergonomics in ERCP? A comparative, simulation-based pilot study. Endosc Int Open. 2024 Mar 18;12(3):E419-E427. doi: 10.1055/a-2231-7393. eCollection 2024 Mar. PMID 38504744
- [Background] Bang JY, Sutton B, Hawes R, Varadarajulu S. Concept of disposable duodenoscope: at what cost? Gut. 2019 Nov;68(11):1915-1917. doi: 10.1136/gutjnl-2019-318227. Epub 2019 Feb 12. No abstract available. PMID 30772837
- [Background] Larsen S, Kalloo A, Hutfless S. The hidden cost of colonoscopy including cost of reprocessing and infection rate: the implications for disposable colonoscopes. Gut. 2020 Feb;69(2):197-200. doi: 10.1136/gutjnl-2019-319108. Epub 2019 Aug 14. No abstract available. PMID 31413166
- [Background] Deb A, Perisetti A, Goyal H, Aloysius MM, Sachdeva S, Dahiya D, Sharma N, Thosani N. Gastrointestinal Endoscopy-Associated Infections: Update on an Emerging Issue. Dig Dis Sci. 2022 May;67(5):1718-1732. doi: 10.1007/s10620-022-07441-8. Epub 2022 Mar 9. PMID 35262904
- [Background] Barakat MT, Banerjee S. Novel Algorithms for Reprocessing, Drying and Storing Endoscopes. Gastrointest Endosc Clin N Am. 2020 Oct;30(4):677-691. doi: 10.1016/j.giec.2020.06.003. Epub 2020 Jul 30. PMID 32891225
- [Background] Han ZL, Lin BT, Wang ZJ, Chen X, Xi YY, Wang JF, Qiao WG, Huang Y, Lin ZZ, Huang SH, Chua TY, Liu SD, Luo XB. Evaluation of a novel disposable esophagogastroduodenoscopy system in emergency, bedside, and intraoperative settings: Pilot study (with videos). Dig Endosc. 2023 Nov;35(7):857-865. doi: 10.1111/den.14548. Epub 2023 Apr 5. PMID 36905288
- [Background] Ebigbo A, Tadic V, Schlottmann J, Braun G, Prinz F, Wanzl J, Ayoub M, Kraus L, Scheppach M, Nagl S, Schnoy E, Weber T, Probst A, Messmann H, Rommele C. Evaluation of a single-use gastroscope in patients presenting with suspected upper gastrointestinal hemorrhage: a pilot feasibility study (One-Scope I). Endoscopy. 2023 Oct;55(10):940-944. doi: 10.1055/a-2089-5969. Epub 2023 May 9. PMID 37160261
- [Background] van der Ploeg K, de Jonge PJF, Lammers WJ, Koch AD, Vos MC, Paulsen V, Aabakken L, Bruno M. Performance of a single-use gastroscope for esophagogastroduodenoscopy: Prospective evaluation. Endosc Int Open. 2024 Mar 18;12(3):E428-E434. doi: 10.1055/a-2271-2303. eCollection 2024 Mar. PMID 38504741
- [Background] Li DF, Shi RY, Tian YH, Xu ZL, Zhou YS, Sun XJ, Cai JW, Fang YY, Peng H, Wang JM, Dong T, Cai YD, Yao J, Wang LS. The feasibility and safety of disposable endoscope vs. conventional endoscope for upper gastrointestinal tract examination: a multicenter, randomized, parallel, non-inferiority trial. Z Gastroenterol. 2022 Sep;60(9):1314-1319. doi: 10.1055/a-1555-0568. Epub 2021 Nov 12. PMID 34768288
- [Background] Luo X, Ji M, Zhang S, Chen X, Zong Y, Zhang X, Hu H, Hao X, Shao L, Sun C, Shi H, Wang J, Wang B, Li P. Disposable versus reusable gastroscopes: a prospective randomized noninferiority trial. Gastrointest Endosc. 2022 Aug;96(2):250-261. doi: 10.1016/j.gie.2022.03.024. Epub 2022 Apr 4. PMID 35381230
- [Background] Ramai D, Smit E, Kani HT, Papaefthymiou A, Warner L, Chandan S, Dhindsa B, Facciorusso A, Gkolfakis P, Ofosu A, Barakat M, Adler DG. Cannulation rates and technical performance evaluation of commericially available single-use duodenoscopes for endoscopic retrograde cholangiopancreatography: A systematic review and meta-analysis. Dig Liver Dis. 2024 Jan;56(1):123-129. doi: 10.1016/j.dld.2023.02.022. Epub 2023 Mar 30. PMID 37003844
- [Background] Bruno MJ, Beyna T, Carr-Locke D, Chahal P, Costamagna G, Devereaux B, Giovannini M, Goenka MK, Khor C, Lau J, May G, Muthusamy VR, Patel S, Petersen BT, Pleskow DK, Raijman I, Reddy DN, Repici A, Ross AS, Sejpal DV, Sherman S, Siddiqui UD, Ziady C, Peetermans JA, Rousseau MJ, Slivka A; EXALT Single-use Duodenoscope Study Group. Global prospective case series of ERCPs using a single-use duodenoscope. Endoscopy. 2023 Dec;55(12):1103-1114. doi: 10.1055/a-2131-7180. Epub 2023 Jul 18. PMID 37463599
- [Background] Ross AS, Bruno MJ, Kozarek RA, Petersen BT, Pleskow DK, Sejpal DV, Slivka A, Moore D, Panduro K, Peetermans JA, Insull J, Rousseau MJ, Tirrell GP, Muthusamy VR. Novel single-use duodenoscope compared with 3 models of reusable duodenoscopes for ERCP: a randomized bench-model comparison. Gastrointest Endosc. 2020 Feb;91(2):396-403. doi: 10.1016/j.gie.2019.08.032. Epub 2019 Nov 1. PMID 31679738
- [Background] Forbes N, Elmunzer BJ, Allain T, Parkins MD, Sheth PM, Waddell BJ, Du K, Douchant K, Oladipo O, Saleem A, Cartwright S, Chau M, Howarth M, McKay J, Nashad T, Ruan Y, Bishay K, Gonzalez-Moreno E, Meng ZW, Bass S, Bechara R, Cole MJ, Jalink DW, Mohamed R, Turbide C, Belletrutti PJ, Kayal A, Kumar PR, Hilsden RJ, Buret AG, Hookey L, Heitman SJ. Effect of Disposable Elevator Cap Duodenoscopes on Persistent Microbial Contamination and Technical Performance of Endoscopic Retrograde Cholangiopancreatography: The ICECAP Randomized Clinical Trial. JAMA Intern Med. 2023 Mar 1;183(3):191-200. doi: 10.1001/jamainternmed.2022.6394. PMID 36689215
- [Background] Turk DJ, Kozarek RA, Botoman VA, Patterson DJ, Ball TJ. Disposable endoscopic biopsy forceps: comparison with standard forceps of sample size and adequacy of specimen. J Clin Gastroenterol. 1991 Feb;13(1):76-8. PMID 2007750
- [Background] Gralnek IM, Stanley AJ, Morris AJ, Camus M, Lau J, Lanas A, Laursen SB, Radaelli F, Papanikolaou IS, Curdia Goncalves T, Dinis-Ribeiro M, Awadie H, Braun G, de Groot N, Udd M, Sanchez-Yague A, Neeman Z, van Hooft JE. Endoscopic diagnosis and management of nonvariceal upper gastrointestinal hemorrhage (NVUGIH): European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2021. Endoscopy. 2021 Mar;53(3):300-332. doi: 10.1055/a-1369-5274. Epub 2021 Feb 10. PMID 33567467
- See also: FDA Continues Efforts to Support Innovation in Medical Device Sterilization — https://www.prnewswire.com/news-releases/fda-continues-efforts-to-support-innovation-in-medical-device-sterilization-301599169.html